

Add contact details of the local research team and either the Chief or Local Investigator

## **CONSENT FORM**

## STEDI: Simulation Training for Emergency Department Imaging (Phase 2)

Chief Investigator: Dr Alex Novak

If you agree, please initial box

| I confirm that I have read the information sheet dated (version) for this study. I have had the opportunity to consider the | | |
|---|---|---|
| information, ask questions and have had these answered satisfactorily. | | |
| I understand that my participa any time without giving any re | • | |
| 3. I understand that data collected of Oxford University Hospitals NHS the local NHS Trust, where it is repermission for these individuals to | FT (as sponsor), from reg<br>elevant to my taking part ir | ulatory authorities or from<br>n this research. I give |
| I understand who will have ac be stored and what will happe | • | |
| 5. I understand that the information other research in the future, and | | |
| 6. I understand how to raise a co | oncern or make a compl | aint. |
| 7. I agree to take part in this stud | dy. | |
| Name of Participant | Date | Signature |
| Name of Person taking consent | | Signature |
| 1copy for participant; 1 copy for researcher site | | |
| | Version 1.0 28-Mar-2022<br>Department Imaging (Ph | ase 2) IRAS Project number: < > |

Chief Investigator: Dr Alex Novak

REC Ref:R80145/RE001 Page: 1 of 1